CLINICAL TRIAL: NCT05025397
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Danavorexton in Anesthetized Adults
Brief Title: A Study of Danavorexton in Anesthetized Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: TAK-925-1019
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-925; Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1: Danavorexton Low Dose (Experimental): Danavorexton low dose or danavorexton placebo-matching infusion, once, intravenously on Day 1 in healthy adult participants with intravenous propofol as induction anesthetic and inhaled sevoflurane as the primary maintenance anesthetic.
  Interventions: Drug: Danavorexton; Drug: Danavorexton Placebo; Drug: Propofol; Drug: Sevoflurane
- Cohort A2: Danavorexton Middle Dose (Experimental): Danavorexton middle dose or danavorexton placebo-matching infusion, once, intravenously on Day 1 in healthy adult participants with intravenous propofol as induction anesthetic and inhaled sevoflurane as the primary maintenance anesthetic.
  Interventions: Drug: Danavorexton; Drug: Danavorexton Placebo; Drug: Propofol; Drug: Sevoflurane
- Cohort A3: Danavorexton High Dose (Experimental): Danavorexton high dose or danavorexton placebo-matching infusion, single, intravenously on Day 1 in healthy adult participants with intravenous propofol as induction anesthetic and inhaled sevoflurane as the primary maintenance anesthetic.
  Interventions: Drug: Danavorexton; Drug: Danavorexton Placebo; Drug: Propofol; Drug: Sevoflurane
- Cohort P: Danavorexton TBD (Experimental): Danavorexton dose to be decided (TBD) or danavorexton placebo-matching infusion, once, intravenously on Day 1 in healthy adult participants with intravenous propofol as induction and primary maintenance anesthetic.
  Dose of danavorexton will be based on the review of observed safety and tolerability data and pharmacokinetic (PK) data of previous cohorts.
  Interventions: Drug: Danavorexton; Drug: Danavorexton Placebo; Drug: Propofol

INTERVENTIONS:
Drug: Danavorexton — Danavorexton intravenous infusion.
  Other Names: TAK-925
Drug: Danavorexton Placebo — Danavorexton placebo-matching intravenous infusion.
Drug: Propofol — Propofol intravenous bolus.
  Arms: Cohort A1: Danavorexton Low Dose; Cohort A2: Danavorexton Middle Dose; Cohort A3: Danavorexton High Dose
Drug: Sevoflurane — Sevoflurane inhalation.
  Arms: Cohort A1: Danavorexton Low Dose; Cohort A2: Danavorexton Middle Dose; Cohort A3: Danavorexton High Dose
Drug: Propofol — Propofol intravenous infusion.
  Arms: Cohort P: Danavorexton TBD

SUMMARY:
The aims of the study are:

* to assess the safety profile of danavorexton when it is administered with anesthetics.
* to learn what effect danavorexton has on anesthetized adults.

On Day 1, participants will receive a single intravenous (IV) infusion of danavorexton or a placebo after participants have been anesthetized for about 40 minutes. Clinic doctors will arrange a follow-up visit by phone or video on Day 7.

DETAILED DESCRIPTION:
The drug being tested in this study is called danavorexton or TAK-925. Danavorexton is being tested to evaluate safety, tolerability, PK, and pharmacodynamics (PD) in healthy participants.

The study will enroll approximately 28 participants. This study consists of 4 cohorts: Cohorts A1, A2, A3 and P (healthy participants aged 18 to 55 years). In each of the 4 cohorts, participants will be randomly assigned (by chance) to receive danavorexton or danavorexton placebo-matching -which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Cohort A1: Danavorexton Low Dose
* Cohort A2: Danavorexton Middle Dose
* Cohort A3: Danavorexton High Dose
* Cohort P: Danavorexton TBD

Additional optional cohorts may be added to the study based on the outcomes from the mandatory cohorts described above.

This trial will be conducted in the United States. The overall time to participate in this study is 37 days including screening period, residential period, and safety follow up period. A follow-up visit by phone or video will be conducted on Day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Current non-smoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months before the administration of the study drug.
2. Has regular sleep-wake habits (example, routinely spends 6.5 to 9 hours in bed nightly).
3. Aged 18 to 55 years, inclusive, at the screening visit.
4. Has a body mass index (BMI) greater than or equal to (>=) 18 and less than or equal to (<=) 32 kilogram per square meter (kg/m^2) at the screening visit.
5. Must be American Society of Anesthesiologists (ASA) Classification I with a Mallampati score less than (<) III, and judged to be in good health based on results of safety laboratory tests (biochemistry, hematology, and urinalysis testing) performed at the screening visit and on medical history, physical examination, vital-sign measurements, and 12-lead electrocardiogram (ECG) performed at screening and Study Day 1 visits.
6. Not expected to have difficulty with the use of an laryngeal mask airway (LMA) as determined by the anesthesiologist or site staff.

Exclusion Criteria:

1. Received immunotherapy within the past year.
2. Has a history or family history of malignant hyperthermia or are known or suspected to have an allergy to inhalational anesthetics, propofol, neuromuscular blocking agents and/or other drugs used during general anesthesia.
3. Has facial hair that could interfere with the seal of a facemask per investigator or site staff and is unwilling to shave it off before check-in.
4. Has undergone major surgery or donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 4 weeks before the screening visit.
5. Has a risk of suicide according to endorsement of Item 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at the screening/baseline visit or have made a suicide attempt in the previous 6 months.
6. Has a positive alcohol or drug screen at screening or Day 1 or has a history of alcohol consumption exceeding 2 standard drinks per day on average within the 12 months before screening. Participants who test positive for cannabis will be excluded.
7. Has caffeine consumption of more than 400 milligram per day (mg/day) for 2 weeks before screening (1 serving of coffee is approximately equivalent to 120 milligram [mg] of caffeine).
8. Has a screening ECG with a QT interval with Fridericia correction method (QTcF) greater than (>) 450 millisecond (ms) (men) or >470 ms (women).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants With at Least one Treatment-emergent Adverse Event (TEAE) | Up to Day 7

SECONDARY OUTCOMES:
Ceoi: Observed Plasma Concentration at the end of Infusion for Danavorexton | Day 1: Pre-anesthesia, pre-infusion and at multiple timepoints (up to 24 hours) post-infusion
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Danavorexton | Day 1: Pre-anesthesia, pre-infusion and at multiple timepoints (up to 24 hours) post-infusion
AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Danavorexton | Day 1: Pre-anesthesia, pre-infusion and at multiple timepoints (up to 24 hours) post-infusion

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Endeavor Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61421bb6c15195002c0ba2d8